CLINICAL TRIAL: NCT03072121
Title: Study of Curative Effect Evaluation of Shexiang Baoxin Pill on Coronary Artery Disease Not Amenable to Revascularization on the Basis of Western Medicine Therapy
Brief Title: Curative Effect Evaluation of Shexiang Baoxin Pill on Coronary Artery Disease Not Amenable to Revascularization
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jun Li (Other)
Collaborators: Shanghai Hutchison Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor-Investigator, Jun Li, Director of Cardiology, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SBP-2016
Record Dates: First submitted 2017-02-22; First posted 2017-03-07 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Coronary Artery Disease(CAD)
Keywords: coronary artery disease; revascularization; Shexiang Baoxin Pill
MeSH Terms: conditions — Coronary Artery Disease | interventions — shexiang baoxin; Clopidogrel; Tablets; Atorvastatin; isosorbide-5-mononitrate; Metoprolol; Trimetazidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shexiang baoxin pill (Experimental): Shexiang baoxin 22.5mg pill by mouth,2 pills three times daily for 6 months & Conventional western medicine (including Aspirin Enteric-coated Tablets, Clopidogrel Hydrogen Sulfate 75 MG Oral Tablet, Atorvastatin Calcium, Isosorbide Mononitrate Tab 20 MG, Metoprolol Tartrate Tab 25 MG, Trimetazidine Dihydrochloride Tablets)
  Interventions: Drug: Shexiang Baoxin pill; Drug: Aspirin Enteric-coated Tablets; Drug: Clopidogrel Hydrogen Sulfate 75 MG Oral Tablet; Drug: Atorvastatin Calcium; Drug: Isosorbide Mononitrate Tab 20 MG; Drug: Metoprolol Tartrate Tab 25 MG; Drug: Trimetazidine Dihydrochloride Tablets
- SBP placebo (Placebo Comparator): Placebo shexiang baoxin 22.5mg pill by mouth,2 pills three times daily for 6 months & Conventional western medicine (including Aspirin Enteric-coated Tablets, Clopidogrel Hydrogen Sulfate 75 MG Oral Tablet, Atorvastatin Calcium, Isosorbide Mononitrate Tab 20 MG, Metoprolol Tartrate Tab 25 MG, Trimetazidine Dihydrochloride Tablets)
  Interventions: Drug: SBP placebo; Drug: Aspirin Enteric-coated Tablets; Drug: Clopidogrel Hydrogen Sulfate 75 MG Oral Tablet; Drug: Atorvastatin Calcium; Drug: Isosorbide Mononitrate Tab 20 MG; Drug: Metoprolol Tartrate Tab 25 MG; Drug: Trimetazidine Dihydrochloride Tablets

INTERVENTIONS:
Drug: Shexiang Baoxin pill — Conventional western medicine & shexiang baoxin pill
  Other Names: SBP
  Arms: Shexiang baoxin pill
Drug: SBP placebo — Conventional western medicine & placebo (for shexiang baoxin pill)
  Arms: SBP placebo
Drug: Aspirin Enteric-coated Tablets — 100mg tablet, one tablet daily.
Drug: Clopidogrel Hydrogen Sulfate 75 MG Oral Tablet — one tablet daily. (for patients who can't use aspirin)
  Other Names: Plavix
Drug: Atorvastatin Calcium — 10 mg tablet, two tablets each night.
  Other Names: Lipitor
Drug: Isosorbide Mononitrate Tab 20 MG — 1 tablet two times daily.
  Other Names: Xinkang
Drug: Metoprolol Tartrate Tab 25 MG — 12.5 mg or 25 mg two times daily.
  Other Names: Metoprolol
Drug: Trimetazidine Dihydrochloride Tablets — 20 mg tablet, one tablet three times daily.
  Other Names: Vasorel

SUMMARY:
The purpose of this study is to determine whether Shexiang Baoxin Pill is effective in the treatment of coronary artery disease not amenable to revascularization on the basis of western medicine therapy.

DETAILED DESCRIPTION:
The western medicine treatment for CAD not amenable to revascularization is limited. Shexiang Baoxin Pill, a kind of Chinese patent medicine has been used for treating coronary artery disease in clinical practice in China for many years.

Shexiang baoxin pill(SBP) is applicable to "Qi deficiency and blood stasis syndrome" in traditional Chinese medicine. Recent experimental research has indicated that SBP can improve myocardial ischemia and promote therapeutic angiogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Participants are aged between 45 and 75 years, diagnosed with sever CAD through coronary arteriography which shows that the left main coronary artery and three-vessel have sever diffuse stenosis, calcification or vascular ectasia, be in accordance with Traditional Chinese Medicine syndrome of "Qi deficiency and blood stasis syndrome" or "phlegm and stasis mu-tual obstruction syndrome".

Exclusion Criteria:

* Patients with severe valvular disease, congenital cardiomyopathy decompensation
* Patients with CAD complicated with severe multiple organ disease such as severe heart failure, severe lung, liver or renal dysfunction, peptic ulcer in active stage, or intracranial hemorrhage
* Patients that use high-dose steroids due to connective tissue disease
* Patients with serious infections
* Patients with malignant tumor
* Patients with hematopoietic diseases
* Pregnant or lactating women.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Mortality | Six months after randomisation
  Death caused by cardiovascular disease

SECONDARY OUTCOMES:
Ejection fraction percentage (EF%) | At baseline (before randomisation), and six months after randomisation.
  One of the Echocardiographic parameters
E/A ratio | At baseline (before randomisation), and six months after randomisation.
  One of the Echocardiographic parameters
C-reactive protein (CRP) | At baseline(before randomisation), and six months after randomisation.
  CRP in μg/L
B-type natriuretic peptide (BNP) | At baseline (before randomisation), and six months after randomisation.
  BNP in pg/mL
Hospital readmission rates | At baseline (before randomisation), and six months after randomisation.
  Hospital readmission rates due to coronary artery disease during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, MD, Study Director — Guang'anmen Hospital of China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zhao D. [Why dentists need to learn the epidemiological status and prevention strategy of coronary heart disease in China]. Zhonghua Kou Qiang Yi Xue Za Zhi. 2016 Jul;51(7):385-6. doi: 10.3760/cma.j.issn.1002-0098.2016.07.001. Chinese. PMID 27480425
- [Result] Zhu H, Luo XP, Wang LJ. [Evaluation on clinical effect of long-term shexiang baoxin pill administration for treatment of coronary heart disease]. Zhongguo Zhong Xi Yi Jie He Za Zhi. 2010 May;30(5):474-7. Chinese. PMID 20681275
- [Result] Zhou Z, Shen W, Yu L, Xu C, Wu Q. A Chinese patent medicine, Shexiang Baoxin Pill, for Non-ST-elevation acute coronary syndromes: A systematic review. J Ethnopharmacol. 2016 Dec 24;194:1130-1139. doi: 10.1016/j.jep.2016.11.024. Epub 2016 Nov 12. PMID 27847338
- [Result] Williams B, Menon M, Satran D, Hayward D, Hodges JS, Burke MN, Johnson RK, Poulose AK, Traverse JH, Henry TD. Patients with coronary artery disease not amenable to traditional revascularization: prevalence and 3-year mortality. Catheter Cardiovasc Interv. 2010 May 1;75(6):886-91. doi: 10.1002/ccd.22431. PMID 20432394
- [Result] Gupta S, Pressman GS, Morris DL, Figueredo VM. Distribution of left ventricular ejection fraction in angina patients with severe coronary artery disease not amenable to revascularization. Coron Artery Dis. 2010 Aug;21(5):278-80. doi: 10.1097/MCA.0b013e32833bdf53. PMID 20531008
- [Result] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Result] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2011;9(8):672-7. doi: 10.1016/j.ijsu.2011.09.004. Epub 2011 Oct 13. No abstract available. PMID 22019563
- [Derived] Tian PP, Li J, Gao J, Li Y. Efficacy and safety of the Shexiang Baoxin Pill for the treatment of coronary artery disease not amenable to revascularisation: study protocol for a randomised, placebo-controlled, double-blinded trial. BMJ Open. 2018 Feb 14;8(2):e018052. doi: 10.1136/bmjopen-2017-018052. PMID 29444778